CLINICAL TRIAL: NCT06092567
Title: Post-operative Sensitivity in Composites Using Bulk-fill vs. Oblique Incremental Placement Technique: a Double-blind, Randomized Trial
Brief Title: Post-operative Sensitivity in Composite Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, NEHAL AMIR, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOD/ERB/2022/04
Record Dates: First submitted 2023-09-30; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Class II Dental Caries; Sensitivity, Tooth
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: In this study, participants allocated in two groups by Consecutive non-random sampling technique
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blinded study in which the participant and the outcome assessor masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Oblique Incremental Placement Techniique) (Experimental): In this interventional group, a Nanohybrid composite resin Nexcomp (Meta Biomed, Korea) was placed using an oblique incremental technique with increments not exceeding 2 mm in thickness.
  Interventions: Procedure: Group A ( Oblique Incremental Placement Technique)
- Group B (Bulk-fill Placement Technique) (Experimental): In this group, a composite Beautifil-Bulk Restorative (SHOFU dental) was utilized for restorative purposes using a bulk-fill technique with a thickness of 4 mm.
  Interventions: Procedure: Group B (Bulk-fill Placement technique)

INTERVENTIONS:
Procedure: Group A ( Oblique Incremental Placement Technique) — In this interventional group, a Nanohybrid composite resin Nexcomp (Meta Biomed, Korea) was placed using an oblique incremental technique with increments not exceeding 2 mm in thickness.
  Arms: Group A (Oblique Incremental Placement Techniique)
Procedure: Group B (Bulk-fill Placement technique) — In this group, a composite Beautifil-Bulk Restorative (SHOFU dental) was utilized for restorative purposes using a bulk-fill technique with a thickness of 4 mm
  Arms: Group B (Bulk-fill Placement Technique)

SUMMARY:
Participants will be divided into groups. In group A, Composite restoration done using oblique incremental technique. In group B, Bulk-fill technique was used. VAS scoring to evaluate the primary outcome at one day, one week and two weeks.

DETAILED DESCRIPTION:
After the approval from ethical research committee, a written informed consent taken. Participants were briefed about the intervention with its associated merits and demerits. The restorative procedures were accomplished under rubber dam isolation using adequate local anesthesia. The principles of minimally intervention and adhesive dentistry were employed. Participants were allocated into two groups. In group A, restorative interventive was performed using Oblique incremental placement while in group B, Bulk-fill technique was used. Post-operative sensitivity was recorded at one day, one week and two week follow up using a Visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age with good general health
* Vital and Periodontally stable teeth
* Class-II primary carious lesions with a cavity depth of 3 to 5 mm
* Established contact with adjacent and opposing natural or prosthetic teeth
* Prior defective restorations in need of replacement (secondary caries, marginal fractures, and marginal staining)

Exclusion Criteria:

* Teeth with a history of spontaneous pain
* Compromised oral health status
* Patients with parafunctional habits or temporomandibular disorders
* Previously endodontically treated teeth or evidence of associated periapical/periodontal pathosis
* Participants with a drug history of using anti-inflammatory, analgesics, or psychotropic medications within the last 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Post-operative sensitivity in composite resin restoration | Two weeks
  Evaluation of post-restorative sensitivity in composite restorations using Visual analogue scale score with scoring from 0 to 10. Score 0 (none), 1 to 3 (mild), 4 to 6 (moderate), and 7 to 10 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Amir, BDS, Principal Investigator — Pakistan Institute of Medical Sciences
Locations (1):
- School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afifi SMH, Haridy MF, Farid MR. Evaluation of Post-Operative Sensitivity of Bulk Fill Resin Composite versus Nano Resin Composite: A Randomized Controlled Clinical Study. Open Access Maced J Med Sci. 2019 Jul 26;7(14):2335-2342. doi: 10.3889/oamjms.2019.656. eCollection 2019 Jul 30. PMID 31592052
- [Background] Tardem C, Albuquerque EG, Lopes LS, Marins SS, Calazans FS, Poubel LA, Barcelos R, Barceleiro MO. Clinical time and postoperative sensitivity after use of bulk-fill (syringe and capsule) vs. incremental filling composites: a randomized clinical trial. Braz Oral Res. 2019 Sep 16;33(0):e089. doi: 10.1590/1807-3107bor-2019.vol33.0089. PMID 31531552